CLINICAL TRIAL: NCT03134547
Title: A Comparison of Postoperative Emergence Agitation by Sevoflurane for Intraoperative Sedation Associated With Caudal Block in Children: Randomised Comparison of Two Dose
Brief Title: A Comparison of Emergence Agitation by Sevoflurane for Intraoperative Sedation Associated With Caudal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Eun Kyung Choi, Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YUMC 2017-04-12
Record Dates: First submitted 2017-04-21; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Emergence Agitation
Keywords: emergence agitation; sevoflurane; children
MeSH Terms: conditions — Emergence Delirium | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low volume volatile anesthetics (Active Comparator): 1.0 % sevoflurane sedation via face mask , low dose sevoflurane group
  Interventions: Drug: low dose sevoflurane group
- high volume volatile anesthetics (Active Comparator): 2.5 % sevoflurane sedation via face mask, high dose sevoflurane group
  Interventions: Drug: high dose sevoflurane group

INTERVENTIONS:
Drug: low dose sevoflurane group — low volume volatile anesthetics (1.0%)
  Other Names: 1.0 %sevoflurane
  Arms: low volume volatile anesthetics
Drug: high dose sevoflurane group — high volume volatile anesthetics (2.5%)
  Other Names: 2.5% sevoflurane
  Arms: high volume volatile anesthetics

SUMMARY:
This study was performed to compare the incidence of EA between two dose of sevoflurane for sedation with caudal block in children, and intended to find the optimal dose for prevention of sevoflurane induced emergence agitation

DETAILED DESCRIPTION:
After approval Institutional Review Board of our institute, informed consent was obtained from the parents of all pediatric patients. 40 children, aged up to 5 yr, undergoing elective subumbilical surgery were enrolled. Children with development delay, anxiety disorder, or a history of allergy to any study drugs, or severe systemic disease were excluded from this study. By a computer generated schedule, children were randomized to either the low dose (1.0%) end tidal concentration of sevoflurane group (Group LS) or the high dose (2.5%) end tidal concentration of sevoflurane group (Group HS). The patients were sedated with intravenous ketamine 2 mg/kg and midazolam 0.05 mg/kg at waiting room and checked the loss of response to verbal or gentle touch. Then the patients were into the operating room, applied electrocardiography (ECG), pulse oximetry, and noninvasive blood pressure. Respiratory rate and end tidal carbon dioxide (CO2) were monitored via face mask. After baseline vital signs were monitored, the patient was posed in lateral Sims position, and 1 ml/kg lidocaine 1% with 5 μg/ml epinephrine was injected into the caudal space using a 22 G needle under 100% oxygen with each sevoflurane concentration according to group through a face mask. All of these procedures were performed by one skilled anesthesiologist who blinded about the study group. After caudal block was performed, the patients were returned in supine position, and maintained on spontaneous ventilation under 100% oxygen and each sevoflurane concentration according to group via face mask to conduct sedation during operation. If oxygen saturation decreases lesser than 90% due to over sedation or breathe holding caused by procedural pain, ventilation was assisted. If analgesia was insufficient for operation, fentanyl 0.5-1 μg/kg was administrated properly.

In the postanesthetic care unit (PACU), the investigators observed EA episodes at 5 and 30 min after PACU arrival using Four-point agitation scale and Pediatric Anesthesia Emergence Delirium (PAED) scale, and if a total score of PAED scale is higher than 15, which is prescribed a severe agitation, and then propofol 0.5 mg/kg was administered. EA was considered as an Four-point agitation scale > 3 or PAED scale > 10.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective subumbilical surgery, American society of anesthesiologist physical status classification 1

Exclusion Criteria:

* Children with development delay, anxiety disorder, or a history of allergy to any study drugs, or severe systemic disease were excluded from this study.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
postoperative agitation score | 5 minutes in the recovery room
  Four-point agitation scale
postoperative agitation score | 30 minutes in the recovery room
  Four-point agitation scale
postoperative agitation score | 5 minutes in the recovery room
  Pediatric Anesthesia Emergence Delirium (PAED) scale
postoperative agitation score | 30 minutes in the recovery room
  Pediatric Anesthesia Emergence Delirium (PAED) scale

CONTACTS AND LOCATIONS:
Overall Officials: Eun kyung Choi, MD,PhD, Principal Investigator — Yeungnam University Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Result] Aono J, Ueda W, Mamiya K, Takimoto E, Manabe M. Greater incidence of delirium during recovery from sevoflurane anesthesia in preschool boys. Anesthesiology. 1997 Dec;87(6):1298-300. doi: 10.1097/00000542-199712000-00006. PMID 9416712